CLINICAL TRIAL: NCT01445730
Title: Fructose Consumption Aggravates Dysregulation of Postprandial Lipid Metabolism in Obese Hypertriglyceridemic Men With High Cardiometabolic Risk Profile and Associates With Liver Fat Deposition
Brief Title: Fructose Consumption and Metabolic Dysregulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marja-Riitta Taskinen (Other)
Collaborators: Sahlgrenska University Hospital (Other); Lund University (Other); University of Naples (Other); Laval University (Other)
Responsible Party: Sponsor-Investigator, Marja-Riitta Taskinen, Professor, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: T1010K0029
Record Dates: First submitted 2011-09-28; First posted 2011-10-04 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Central Obesity; Hypertriglyceridemia
Keywords: fructose; hypertriglyceridemia; postprandial lipids; de novo lipogenesis; stable isotopes
MeSH Terms: conditions — Obesity, Abdominal; Hypertriglyceridemia | interventions — Fructose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- After fructose feeding (Experimental): After 3 month fructose diet 75 g/day
  Interventions: Dietary Supplement: Fructose

INTERVENTIONS:
Dietary Supplement: Fructose — 3 month fructose diet 75 g/day

SUMMARY:
High fructose intake is increasingly recognized as causative in development of prediabetes, metabolic syndrome and cardiovascular disease (CVD). The mechanisms underlying fructose-induced metabolic disturbances are unclear but are beginning to be unraveled. In contrast to metabolism of glucose, the breakdown of fructose leads to the generation of metabolites that stimulate hepatic de novo lipogenesis (DNL) and increased levels of both fasting and postprandial triglycerides. The key lipogenic transcription factor seems to be activated by fructose independently of insulin. However, it is still controversial whether fructose consumption increases DNL in man to the extent that it induces metabolic disturbances. Animal studies have shown that also the adipose tissue is responsive to fructose feeding fructose, and that high fructose-feeding induces insulin resistance and inflammation in the adipose tissue. The role of intestinal insulin resistance in fructose-induced dysmetabolism has not been studied in detail. The critical question is whether the metabolic disturbances are induced by calorie excess or by fructose per se.

DETAILED DESCRIPTION:
Detailed description: Study subjects will participate to studies 1-4 before and 3 m after fructose diet:

1. An oral fat load or a kinetic study with stable isotopes combined with an oral fat load.
2. Determination of liver, subcutaneous and intra-abdominal fat. (Proton magnetic resonance spectroscopy )
3. Lipolytic enzymes, advanced lipid analysis, fat biopsies and genetic studies and gut microbiota profiling
4. Oral glucose tolerance test and analysis of incretins and inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 27-40
* Waist > 96 cm
* Age 20-60 years
* Male

Exclusion Criteria:

* Smoking
* Active health problems
* Contraindications to MRI scanning
* Bleeding tendency
* Abnormal liver or renal function tests
* Type 2 diabetes
* Evidence of metabolic or viral liver disease
* Alcohol intake > 21 units per week
* Chronic medication except ones needed for stable hypertension

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2011-08; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marja-Riitta Taskinen, Professor, Principal Investigator — Helsinki University Central Hospital, Biomedicum
Locations (4):
- Université Laval, Québec, Canada
- Helsinki University Central Hospital, Biomedicum, Helsinki, Finland
- University of Naples, Federico II, and Faculty of Medicine, Naples, Italy
- Sahlgrenska Academy at University of Gothenburg and Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Taskinen MR, Bjornson E, Matikainen N, Soderlund S, Ramo J, Ainola MM, Hakkarainen A, Sihlbom C, Thorsell A, Andersson L, Bergh PO, Henricsson M, Romeo S, Adiels M, Ripatti S, Laakso M, Packard CJ, Boren J. Postprandial metabolism of apolipoproteins B48, B100, C-III, and E in humans with APOC3 loss-of-function mutations. JCI Insight. 2022 Oct 10;7(19):e160607. doi: 10.1172/jci.insight.160607. PMID 36040803

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | After Fructose Feeding
Started | 82
Completed | 71
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — For the advice of a dentist | 1
Not completed — The data from magnetic resonance examinations were not sufficient | 9

BASELINE CHARACTERISTICS:
Population: Of the 82 subjects, two subjects discontinued the intervention study: one developed a skin rash, which was considered as possible allergic reaction to flavouring and the other subject discontinued in response to his dentist's advice. In addition, the data from magnetic resonance examinations at baseline or after the fructose intervention were not sufficient from nine subjects for technical reasons to allow the analyses of different fat depots. Thus, 71 subjects completed the full study protocol.
Arm/Group | After Fructose Feeding
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 82
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 4
  Sweden | 10
  Finland | 50
  Italy | 18

OUTCOME MEASURES:

1. Primary Outcome: TG Plasma AUC
Description: Before vs. after fructose challenge: Triglycerides (TG) plasma Area Under Curve (AUC)
Time Frame: Form the baseline (time point 1) to end of treatment at 3 months (time point 2)
Measure: Mean (Standard Deviation); unit: mmol/l*min
Arm/Group | After Fructose Feeding
Number analyzed (Participants) | 71
mmol/l*min
  Time point 1 | 1130 (590)
  Time point 2 | 1220 (598)
Statistical Analysis 1: Comparison: After Fructose Feeding; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)

2. Primary Outcome: B48 Plasma AUC
Description: Before vs. after fructose challenge: apolipoprotein (apo)B48 plasma Area Under Curve (AUC)
Time Frame: Form the baseline (time point 1) to end of treatment at 3 months (time point 2)
Measure: Mean (Standard Deviation); unit: mg/l*min
Arm/Group | After Fructose Feeding
Number analyzed (Participants) | 71
mg/l*min
  Time point 1 | 7660 (3210)
  Time point 2 | 8200 (3340)
Statistical Analysis 1: Comparison: After Fructose Feeding; Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)

3. Primary Outcome: TG Plasma iAUC
Description: Before vs. after fructose challenge:Triglycerides (TG) plasma incremental Area Under Curve (iAUC)
Time Frame: Form the baseline (time point 1) to end of treatment at 3 months (time point 2)
Measure: Mean (Standard Deviation); unit: mmol/l*min
Arm/Group | After Fructose Feeding
Number analyzed (Participants) | 71
mmol/l*min
  Time point 1 | 377 (422)
  Time point 2 | 422 (270)
Statistical Analysis 1: Comparison: After Fructose Feeding; Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: DNL
Description: Before vs. after fructose challenge: de novo lipogenesis (DNL)
Time Frame: Form the baseline (time point 1) to end of treatment at 3 months (time point 2)
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | After Fructose Feeding
Number analyzed (Participants) | 71
μmol/L
  Time point 1 | 12.3 (10)
  Time point 2 | 16.5 (11)
Statistical Analysis 1: Comparison: After Fructose Feeding; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: ApoC-III
Description: Before vs. after fructose challenge: Apolipoprotein C-III (ApoC-III)
Time Frame: Form the baseline (time point 1) to end of treatment at 3 months (time point 2)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | After Fructose Feeding
Number analyzed (Participants) | 71
mg/dL
  Time point 1 | 10.4 (5.1)
  Time point 2 | 11.2 (5)
Statistical Analysis 1: Comparison: After Fructose Feeding; Test type: Other; p = 0.006, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: β-OH Butyrate
Description: Before vs. after fructose challenge: beta-OH butyrate (β-OH butyrate)
Time Frame: Form the baseline (time point 1) to end of treatment at 3 months (time point 2)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | After Fructose Feeding
Number analyzed (Participants) | 71
mg/dL
  Time point 1 | 0.699 (0.55)
  Time point 2 | 0.542 (0.48)
Statistical Analysis 1: Comparison: After Fructose Feeding; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Liver Fat
Description: Before vs. after fructose challenge
Time Frame: Form the baseline (time point 1) to end of treatment at 3 months (time point 2)
Measure: Mean (Standard Deviation); unit: percentage of liver fat content
Arm/Group | After Fructose Feeding
Number analyzed (Participants) | 71
percentage of liver fat content
  Time point 1 | 6.66 (6.1)
  Time point 2 | 7.33 (6.6)
Statistical Analysis 1: Comparison: After Fructose Feeding; Test type: Other; p = 0.008, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During 3 month fructose diet 75 g/day.
Description: Of the 82 subjects, two subjects discontinued the intervention study: one developed a skin rash, which was considered as possible allergic reaction to flavouring and the other subject discontinued in response to his dentist's advice. In addition, the data from magnetic resonance examinations at baseline or after the fructose intervention were not sufficient from nine subjects for technical reasons to allow the analyses of different fat depots. Thus, 71 subjects completed the full study protocol.
Arm/Group | After Fructose Feeding
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 1/82
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | After Fructose Feeding (N=82)
skin rash (Skin and subcutaneous tissue disorders) | 1 (1) — One subject developed a skin rash which was considered as possible allergic reaction to flavouring. The rash disappeared after the discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2013-08-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT01445730/Prot_000.pdf